CLINICAL TRIAL: NCT06424977
Title: Safety and Effectiveness of Biomarker Targeted Stimulation in Epilepsy
Brief Title: Biomarker Targeted Stimulation for Epileptiform Events
Acronym: BTSEE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cadence Neuroscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAD2004
Record Dates: First submitted 2024-05-09; First posted 2024-05-22 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Biomarker Targeted Stimulation (BTS)

INTERVENTIONS:
Device: Biomarker Targeted Stimulation (BTS) — Using continuous stimulation to target multiple network nodes, Biomarker Targeted Stimulation (BTS) is intended to suppress abnormal interictal activity, as determined by biomarkers including interictal epileptiform discharges (IED) and high frequency oscillations (HFO), with the intention to reduce brain hyperexcitability, thereby limiting seizure occurrence.

SUMMARY:
This is a multicenter, prospective, controlled study designed to evaluate treatment with the BTS System.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 7 years of age.
2. Subject has focal onset seizures.
3. Subject has failed treatment with a minimum of two AED's used in typical therapeutic dosages.
4. Subject has seizures that are distinct, stereotypical events that can be reliably counted by the patient or caregiver.
5. Subject can reasonably be expected to maintain a seizure diary and the BTS System alone, or with the assistance of a competent individual.
6. For one month prior to enrollment, subject's anti-epileptic medication dosages and ketogenic diet (as applicable) have been stable (other than acute, intermittent use of benzodiazepines) and subject has had at least three primary, disabling seizures per month, on average. Seizures must be separated by a minimum of eight hours not to be considered part of a cluster. A cluster, for the purpose of this criterion, shall be considered a single seizure.
7. Subject is able to complete regular office visits and telephone appointments in accordance with the study protocol requirements.
8. A female subject of childbearing age must have a negative serum pregnancy test within two weeks prior to implant of the INSR, and, if sexually active, must be using a reliable form of birth control, be surgically sterile, or be at least two years post-menopausal.
9. Subject has been informed of their eligibility for resective surgery as a potential alternative to the study, if such surgery is a reasonable option.
10. Subject has had a brain MRI epilepsy evaluation within the past two years.
11. Subject's anatomy will permit implantation of the INSR within 20 mm of the skin surface.

Exclusion Criteria:

1. Subject has a history of substance abuse within the preceding two years.
2. Subject participated in another drug or device trial that may confound study results within the preceding 30 days.
3. Subject is implanted with pacemaker, implantable cardiac defibrillator, cardiac management product, or a medical device that interferes with the BTS System or with which the BTS System interferes. Patients with a vagus nerve stimulator (VNS) implanted may be enrolled, provided their clinical status has been stable for at least one month prior to enrollment at their current stimulation parameter settings.
4. Subject has anatomy that may interfere with electrode placement.
5. Subject is on anticoagulants and is unable to discontinue them perisurgically, as required by the neurosurgeon or Investigator.
6. Subject has significant platelet dysfunction from medical conditions or medications (including, particularly, aspirin or sodium valproate). If platelet dysfunction is suspected, subject can be enrolled only if a hematologist, the Investigator, and the neurosurgeon judge it to be advisable.
7. Subject has been diagnosed with psychogenic or non-epileptic seizures that cannot be distinguished from their epileptogenic events.
8. Subject is ineligible for cranial surgery.

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | Intervals through 7, 12, and 24 months post-implant
  Determine adverse event rate, including adverse device effects and serious adverse events

SECONDARY OUTCOMES:
Seizure frequency | Intervals calculated at 4 to 7 months and through 12 and 24 months post-implant.
  Using seizure diaries, calculate disabling seizure frequency, normalized to months, compared to baseline.
Neurocognitive testing | Evaluated at 7 months, 12 months, and 24 months post-implant.
  Neurocognitive tests, using the NIH Toolbox, including the Flanker Inhibitory Control and Attention Test, Picture Sequence Memory Test, and Picture Vocabulary Test, compared to baseline.
Depression testing | Evaluated at 7 months, 12 months, and 24 months post-implant.
  Patient reported depression evaluation using Child Depression Inventory (CDI) or Beck Depression Inventory (BDI) (depending on age), compared to baseline.
Anxiety testing | Evaluated at 7 months, 12 months, and 24 months post-implant.
  Patient reported anxiety evaluation using Revised Children's Manifest Anxiety Scale (RCMAS-2) or Beck Anxiety Inventory (depending on age), compared to baseline.
Quality of life testing | Evaluated at 7 months, 12 months, and 24 months post-implant.
  Patient reported quality of life evaluation using Quality of Life in Childhood Epilepsy Questionnaire (QOLCE-55), Quality of Life in Epilepsy Inventory for Adolescents (QOLIE-AD-48), or Quality of Life in Epilepsy (QOLIE-31) (depending on age), compared to baseline.
Sleep testing | Evaluated at 7 months, 12 months, and 24 months post-implant.
  Patient reported sleep evaluation using Epworth Sleepiness Scale for Children and Adolescents (ESS-CHAD) or Epworth Sleepiness Scale (ESS) (depending on age), compared to baseline.
Seizure severity testing | Evaluated at 7 months, 12 months, and 24 months post-implant.
  Patient reported seizure severity evaluation using Liverpool Seizure Severity Scale 2.0 (LSSS 2.0), compared to baseline.
Caregiver burden testing | Evaluated at 7 months, 12 months, and 24 months post-implant.
  Caregiver reported burden evaluation using Caregiver Burden Inventory (CBI), compared to baseline.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lundstrom BN, Worrell GA, Stead M, Van Gompel JJ. Chronic subthreshold cortical stimulation: a therapeutic and potentially restorative therapy for focal epilepsy. Expert Rev Neurother. 2017 Jul;17(7):661-666. doi: 10.1080/14737175.2017.1331129. Epub 2017 May 25. PMID 28532252
- [Background] Kerezoudis P, Grewal SS, Stead M, Lundstrom BN, Britton JW, Shin C, Cascino GD, Brinkmann BH, Worrell GA, Van Gompel JJ. Chronic subthreshold cortical stimulation for adult drug-resistant focal epilepsy: safety, feasibility, and technique. J Neurosurg. 2018 Aug;129(2):533-543. doi: 10.3171/2017.5.JNS163134. Epub 2017 Oct 20. PMID 29053073
- [Background] Lundstrom BN, Gompel JV, Khadjevand F, Worrell G, Stead M. Chronic subthreshold cortical stimulation and stimulation-related EEG biomarkers for focal epilepsy. Brain Commun. 2019;1(1):fcz010. doi: 10.1093/braincomms/fcz010. Epub 2019 Sep 6. PMID 31667473
- [Background] Starnes K, Miller K, Wong-Kisiel L, Lundstrom BN. A Review of Neurostimulation for Epilepsy in Pediatrics. Brain Sci. 2019 Oct 18;9(10):283. doi: 10.3390/brainsci9100283. PMID 31635298
- [Background] Alcala-Zermeno JL, Gregg NM, Van Gompel JJ, Stead M, Worrell GA, Lundstrom BN. Cortical and thalamic electrode implant followed by temporary continuous subthreshold stimulation yields long-term seizure freedom: A case report. Epilepsy Behav Rep. 2020 Sep 2;14:100390. doi: 10.1016/j.ebr.2020.100390. eCollection 2020. PMID 32995742